CLINICAL TRIAL: NCT05396248
Title: Use of a Memory Technique to Improve New Learning and Memory in Individuals With Mild Cognitive Impairment
Brief Title: Improve New Learning and Memory in Individuals With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: University of Michigan (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-1183-22
Record Dates: First submitted 2022-05-18; First posted 2022-05-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Memory; learning; rehabilitation; aging; cognition
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive memory retraining exercises administered on a laptop computer twice a week for five weeks (10 training sessions).
  Interventions: Behavioral: Memory Retraining Exercises
- Placebo Control Group (Placebo Comparator): The placebo control group will receive placebo memory exercises administered on a laptop computer twice a week for five weeks (10 placebo control sessions).
  Interventions: Behavioral: Placebo Control Memory Exercises

INTERVENTIONS:
Behavioral: Memory Retraining Exercises — Memory retraining exercises will be administered on a laptop computer twice a week for five weeks (10 training sessions).
  Arms: Experimental Group
Behavioral: Placebo Control Memory Exercises — Placebo control memory exercises will be administered on a laptop computer twice a week for five weeks (10 training sessions).
  Arms: Placebo Control Group

SUMMARY:
The current study is a double-blind, placebo-control randomized clinical trial examining the efficacy of memory retraining in individuals with Mild Cognitive Impairment (MCI). Impairment in higher level cognitive processing, such as new learning and memory, is one of the most common deficits in individuals with MCI and such deficits have been shown to exert significant negative impact on multiple aspects of everyday life, including occupational and social functioning. Despite these findings, few studies have attempted to treat these cognitive deficits in order to improve the everyday functioning of individuals with MCI. Through a small randomized clinical trial, the investigators found that individuals with MCI with documented cognitive impairment show a significant improvement in their memory performance following a treatment protocol designed to facilitate learning. The current proposal will replicate this finding and further evaluate (a) the impact of the treatment on everyday functioning, (b) the long term efficacy of the treatment and (c) the utility of booster sessions in facilitating long-term treatment effects. We will randomly assign older individuals who meet criteria for a diagnosis of amnestic MCI to a memory retraining group or a placebo control group. Both groups will undergo baseline, immediate and long-term follow-up assessment consisting of: (1) a traditional neuropsychological battery, (2) an assessment of global functioning examining the impact of the treatment on daily activities, and (3) functional neuroimaging. This design will allow the investigators to evaluate the efficacy of this particular memory retraining technique in an aMCI population through the assessment of cognitive function via a standard evaluation. In addition, the investigators will be able to draw conclusions regarding the impact of this particular memory remediation program on everyday life from questionnaires completed by the participant and a significant other. Optional enrollment in pre- post neuroimaging will also allow the investigators to look at changes in the brain.

ELIGIBILITY:
Inclusion Criteria:

* 60 or older.
* read and speak English fluently.
* Research based diagnosis of Amnestic Mild Cognitive Impairment

Exclusion Criteria:

* prior stroke or neurological injury/disease (i.e. traumatic brain injury, Multiple Sclerosis, or Stroke).
* history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis).
* significant alcohol or drug abuse history (inpatient treatment).
* Benzodiazepines and steroid use

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Verbal list learning | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score from Open-Trial Selective Reminding Test (OT-SRT)
Participation in everyday life | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score from Participation Assessment with Recombined Tools

SECONDARY OUTCOMES:
Self-reported depression | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score on the Geriatric Depression Scale
Self-reported anxiety | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score on the Geriatric Anxiety Scale
Self-reported quality of life | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score on the Quality of Life in Alzheimer's Disease
Self-reported quality of well-being | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score on the Quality of Well-Being Scale - Self-Administered
Functional neuroimaging | two points in time: pre-treatment and immediately following treatment
  Change in total scores from memory task during fMRI scan
Functional memory | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score from Object Location Task
Functional memory | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score from the modified Everyday Memory Scenarios (EMS)
Story memory | four points in time: pre-treatment, immediately following treatment, and 6- and 18- months after treatment is completed
  Change in total score from Prose Memory Test

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, Principal Investigator — Kessler Foundation
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Kessler Foundation Research Center, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided